CLINICAL TRIAL: NCT03356041
Title: The Role of a Clinical Pharmacist in Lifestyle Modification
Brief Title: The Role of a Clinical Pharmacist in Lifestyle Modification in Type 2 Diabetic Patients With Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Kawa Dizaye, Professor of Pharmacology, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Hawler Med University
Record Dates: First submitted 2017-11-17; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): The intervention group will receive the three months' lifestyle modification program by a clinical pharmacist.
  Interventions: Other: Diabetic patients with neuropathy
- Usual care Group (No Intervention): The usual care group will be provided the standard medical services

INTERVENTIONS:
Other: Diabetic patients with neuropathy — Lifestyle modification will be assessed using summary of diabetes self-care activity
  Other Names: Intervention group
  Arms: Intervention Group

SUMMARY:
The aims of this study are to determine the prevalence of diabetic peripheral neuropathy among the diabetic patients, to determine the association between the clinical profiles of the diabetic patients (diabetes type, diabetes duration, HbA1c, body mass index, hypertension, total cholesterol) and the diabetic peripheral neuropathy DPN and the rational poly pharmacy used to control pain.

ELIGIBILITY:
Inclusion criteria

1. Aged 18 years or older.
2. Both sex.
3. Diagnosed with type 2 diabetes at least one year previously.
4. Took at least one prescribed medication for diabetes.
5. Diagnosed as diabetic peripheral neuropathy based on clinical

Exclusion Criteria:

1. History of alcohol consumption.
2. Thyroid gland disorder.
3. Any kidney disorder.
4. Any conditions that could confound assessment of pain due to diabetic peripheral neuropathy.
5. Have foot injury or open sore.
6. Pregnant females or who plan to become pregnant during the study period.
7. Any serious medical condition that might prevent completion or hinder compliance with exercise.

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-12-20 (Estimated); Primary Completion 2018-03-16 (Estimated); Study Completion 2018-03-23 (Estimated)

PRIMARY OUTCOMES:
Estimating Summary of diabetes self-care activity (SDSCA) | Three months
  Assessing Lifestyle modification by summary of diabetes self-care activity (SDSCA) at baseline visit and after three months for both Intervention patients and usual care group Increases in the means of the items of the scale as Exercise, Blood sugar testing, Specific diet and Foot care in the intervention group.
Adherence to treatment according to Morisky scale | Three months
  Morisky scale is used to assess medication adherence at baseline visit and after three months for both Intervention patients and usual care group.
  Improving the patient medication adherence behavior in the intervention group patients
Douleur Neuropathique 4 (DN4), Neuropathic Pain Scale (NPS), | Three months
  Reduction in the percent of response of patients feeling; electric shock, tingling, and pin needle after the lifestyle modification in the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Kawa Dizaye, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: Undecided